CLINICAL TRIAL: NCT02344940
Title: Safety of Toremifene and Tamoxifen Therapy in Premenopausal Patients With Operable Breast Cancer: A Randomized, Controlled, Prospective, Observational Study
Brief Title: Safety of Toremifene and Tamoxifen Therapy in Premenopausal Patients With Operable Breast Cancer
Acronym: TTOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1401
Record Dates: First submitted 2015-01-05; First posted 2015-01-26 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: operable; premenopausal; endocrine therapy; safety; tamoxifen; toremifene
MeSH Terms: conditions — Breast Neoplasms | interventions — Toremifene; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- toremifene (Experimental): patients who will be treated with toremifene.
  Interventions: Drug: Toremifene
- tamoxifen (Active Comparator): patients who will be treated with tamoxifen.
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Toremifene — patients will take toremifene 60 mg qd.
  Other Names: Fareston
  Arms: toremifene
Drug: Tamoxifen — patients will take tamoxifen 10 mg bid.
  Arms: tamoxifen

SUMMARY:
To compare the safety of toremifene and tamoxifen therapy in premenopausal patients with operable breast cancer by monitoring gynecological abnormality,blood lipid level,hepatic abnormality,estrogen level and perimenopausal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18 years, premenopausal
2. Histologically confirmed invasive breast cancer by core needle biopsy, hormonal receptor positive, defined as estrogen receptor(ER)/progesterone receptor(PR) positive
3. Patients must have received standard local therapy: normalized modified radical mastectomy or breast conserving surgery with negative margin and post-surgical radiotherapy. Patient should completed adjuvant therapy according to conditions, including adjuvant radiotherapy, neoadjuvant or adjuvant chemotherapy.
4. Leukocyte ≥ 3*109/L; Platelets ≥ 75*109/L; Serum glutamate oxaloacetate(AST/SGOT) or serum glutamic-pyruvic transaminase(ALT/SGPT) <2.5 times of upper limit of normal (UNL) range Serum creatinine/blood urea nitrogen(BUN) ≤ upper limit of normal (UNL) range; Written informed consent according to the local ethics committee requirements.
5. Has Eastern Cooperative Oncology Group(ECOG) Performance Score 0-2;

Exclusion Criteria:

1. Histologically confirmed hormonal receptor negative.
2. Have received neoadjuvant/adjuvant endocrine therapy.
3. With metastatic tumor.
4. Family history of endometrial cancer or ovarian cancer or any other kind of gynecological malignant tumor.
5. Have already been detected of ovarian abnormality or endometrial thickening by transvaginal ultrasound.
6. With any of complications that will increase sex hormone level: pituitary adenoma，ovarian tumor, thymic cancer，etc.
7. With any of complications that will decrease sex hormone level:hyperthyroidism，hypothyroidism，liver cirrhosis，severe malnutrition，Turner's syndrome，sex hormone synthetase deficiency, intracranial tumor, pituitary atrophy, etc.
8. Ovarian ablation or suppression
9. With severe non-malignant co-morbidity that will influence long-term follow up.
10. With severe hepatic dysfunction, Child-Pugh C.
11. With severe cardiac dysfunction, New York Heart Association (NYHA) grading III or worse.
12. Known severe hypersensitivity to any drugs in this study;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-12; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
incidence of ovarian cyst | participants will be followed during the first year of endocrine therapy
  Ovarian cyst is defined as a purely liquid-filled structure that was equal to or exceeded 2 cm in its largest diameter detected by transvaginal ultrasonography.Participants will be required to receive transvaginal ultrasonography every 3 months.

SECONDARY OUTCOMES:
incidence of endometrial thickening | participants will be followed during the first year of endocrine therapy
  Endometrial thickness as measured with transvaginal ultrasonography is equal to or exceeded 8mm.Participants will be required to receive transvaginal ultrasonography every 3 months.
change of female hormones | participants will be followed during the first year of endocrine therapy
  Change of follicle stimulating hormone(FSH),luteinizing hormone(LH),estradiol(E2) as measured every 3 months
change of blood lipid | participants will be followed during the first year of endocrine therapy
  Change of blood lipid as measured every 3 months
change of liver function | participants will be followed during the first year of endocrine therapy
  change of blood lipid as measured every 3 months
incidence of fatty liver | participants will be followed during the first year of endocrine therapy
  Incidence of fatty liver as examined by liver ultrasound every 3 months.
change of Kupperman index | participants will be followed during the first year of endocrine therapy
  change of Kupperman index as measured every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, Professor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Hong J, Huang J, Shen L, Zhu S, Gao W, Wu J, Huang O, He J, Zhu L, Chen W, Li Y, Chen X, Shen K. A prospective, randomized study of Toremifene vs. tamoxifen for the treatment of premenopausal breast cancer: safety and genital symptom analysis. BMC Cancer. 2020 Jul 16;20(1):663. doi: 10.1186/s12885-020-07156-x. PMID 32677982